CLINICAL TRIAL: NCT04061668
Title: Single Path Versus Double Path PECS I and II Blocks as an Efficient Analgesic Choice in Female Breast Surgeries. A Prospective Study
Brief Title: Single Path Versus Double Path PECS I and II Blocks as an Efficient Analgesic Choice in Female Breast Surgeries.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hoda Shokri, Associate professor of Anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU R 04/ 2019
Record Dates: First submitted 2019-08-17; First posted 2019-08-20 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Analgesia
Keywords: PECS; bupivacaine
MeSH Terms: conditions — Agnosia | interventions — Dental Occlusion

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- single needle path PECS I and II block group( (Other): The probe is placed inferior to the clavicle . A probe and needle is introduced with in-plane technique . The US is placed below outer third of the clavicle showing pectoralis major and minor muscles then moved infero-laterally to locate fourth rib where pectoralis major and pectoralis minor muscles is visualised . The US probe is moved toward anterior axillary line till pectoralis minor and serratus anterior muscles will be identified at 4th rib at the level of thoraco-acromial artery then the needle is inserted from caudal to cranial using an inclined manner, 15mL of bupivacaine 0.25% is put between pectoralis minor muscle and serratus muscle (PECS II) then it is withdrawn to inject 15 ml of bupivacaine in thel plane between pectoralis muscles . The block will be performed with needle introduced in-plane with the ultrasound probe, and the local anesthetic injection will be visualized .
  Interventions: Other: single needle path PECS I and II block group
- double needle path PECS I and II block group (Sham Comparator): The probe will be placed below outer third of the clavicle showing pectoralis major and minor muscles and the thoraco- acromial artery then moved inferolaterally to locate fourth rib where pectoralis major and pectoralis minor muscles are visualised, then the needle is inserted in plane with probe and 15mL of bupivacaine are put into between pectoralis muscles. In the second puncture , the US probe is moved toward anterior axillary line till pectoralis minor and serratus anterior muscles are identified , the needle will be inserted in plane with the probe from caudal to cranial , 15mL of bupivacaine will be put into the potential space between pectoralis minor muscle and serratus muscle (PECS II).
  Interventions: Other: double needle path PECS I and II block group

INTERVENTIONS:
Other: single needle path PECS I and II block group — The probe is placed inferior to the clavicle . The US probe is placed below outer third of the clavicle showing pectoralis major and minor muscles and the thoraco- acromial artery then moved infero-laterally to locate fourth rib where pectoralis major and pectoralis minor muscles will be visualised . The probe is moved toward anterior axillary line till pectoralis minor and serratus anterior muscles ise identified at 4th rib at the level of thoraco-acromial artery , the needle is inserted in plane with the probe from caudal to cranial using an inclined manner, 15mL of bupivacaine is put into the potential space between pectoralis minor muscle and serratus muscle (PECS II) then it is withdrawn to inject another 15 ml of bupivacaine in the plane between pectoralis muscles . The block will be performed with needle introduced in-plane with the ultrasound probe, and the local anesthetic injection is visualised.
  Other Names: single needle path PECS I and II block
  Arms: single needle path PECS I and II block group(
Other: double needle path PECS I and II block group — The US probe will be initially placed below outer third of the clavicle after skin sterilization showing pectoralis major and minor muscles and the thoraco- acromial artery then moved inferolaterally to locate fourth rib where pectoralis major and pectoralis minor muscles will be visualised, then the needle will be inserted in plane with the probe and 15mL of bupivacaine 0.25% after negative aspiration will be put into the potential space between pectoralis muscles. In the second puncture , the US probe will be moved toward anterior axillary line till pectoralis minor and serratus anterior muscles will be identified at 4th rib at the level of thoraco-acromial artery then the needle will be inserted in plane with the probe from caudal to cranial in an inclined way, 15mL of bupivacaine 0.25% after negative aspiration will be put into the potential space between pectoralis minor muscle and serratus muscle (PECS II).
  Other Names: double needle path PECS I and II block
  Arms: double needle path PECS I and II block group

SUMMARY:
The patients are allocated by computer generated random number method into 2 groups: single needle path PECS I and II block group, where patients receive induction with pec I and II blocks which are performed under ultrasound guidance , with a linear ultrasound transducer on the same side of surgery. The patients are placed in the supine position where the elbow was flexed and shoulder will be abducted. The probe is placed inferior to the clavicle . A linear probe and a beveled tip needle will be introduced with an in-plane technique . The US probe is initially placed below outer third of the clavicle after skin sterilization showing pectoralis major and minor muscles and the thoraco- acromial artery then moved infero-laterally to locate fourth rib where pectoralis major and pectoralis minor muscles are visualised . The US probe is then moved toward anterior axillary line till pectoralis minor and serratus anterior muscles are identified at 4th rib at the level of thoraco-acromial artery then the needle is inserted in plane with the probe from caudal to cranial using an inclined manner, 15mL of bupivacaine will be put into the potential space between pectoralis minor muscle and serratus muscle (PECS II) then it will be withdrawn to inject another 15 ml of bupivacaine in the plane between pectoralis muscles . The block will be performed with needle introduced in-plane with the ultrasound probe, and the local anesthetic (LA) injection is visualized .

In double needle path PECS I and II block group The probe is initially placed below outer third of the clavicle after skin sterilization showing pectoralis major and minor muscles and the thoraco- acromial artery then moved inferolaterally to locate fourth rib where pectoralis major and pectoralis minor muscles are visualised, then the needle is inserted in plane with the probe and 15mL of bupivacaine is put into the potential space between pectoralis muscles. In the second puncture , the probe is moved toward anterior axillary line till pectoralis minor and serratus anterior muscles will be identified at 4th rib at the level of thoraco-acromial artery then the needle will be inserted in plane with the probe from caudal to cranial , 15mL of bupivacaine is put into the potential space between pectoralis minor muscle and serratus muscle (PECS II).

DETAILED DESCRIPTION:
The patients will be randomly allocated by computer generated random number method into 2 groups: single needle path PECS I and II block group(n = 30) where patients will receive induction with pec I and II blocks which will be performed under ultrasound guidance (S-Nerve; Sono-Site Iberica S.L, Madrid, Spain), with a linear ultrasound transducer(10-12 MHz) on the same side of surgery. The patients will be placed in the supine position where the elbow was flexed and shoulder will be abducted. The probe will be placed inferior to the clavicle . A linear probe and a beveled tip needle will be introduced with an in-plane technique . The US probe will be initially placed below outer third of the clavicle after skin sterilization showing pectoralis major and minor muscles and the thoraco- acromial artery then moved infero-laterally to locate fourth rib where pectoralis major and pectoralis minor muscles will be visualised . The US probe was then moved toward anterior axillary line till pectoralis minor and serratus anterior muscles will be identified at 4th rib at the level of thoraco-acromial artery then the needle will be inserted in plane with the probe from caudal to cranial using an inclined manner, 15mL of bupivacaine 0.25% after negative aspiration will be put into the potential space between pectoralis minor muscle and serratus muscle (PECS II) then it will be withdrawn to inject another 15 ml of bupivacaine 0.25% in the fascial plane between pectoralis muscles . The block will be performed with needle (22-G, 80-mm (SonoTap, Pajunk, Geisingen, Germany) introduced in-plane with the ultrasound probe, and the local anesthetic (LA) injection will be visualized in real-time .

In double needle path PECS I and II block group (n = 30) The US probe will be initially placed below outer third of the clavicle after skin sterilization showing pectoralis major and minor muscles and the thoraco- acromial artery then moved inferolaterally to locate fourth rib where pectoralis major and pectoralis minor muscles will be visualised, then the needle will be inserted in plane with the probe and 15mL of bupivacaine 0.25% after negative aspiration will be put into the potential space between pectoralis muscles. In the second puncture , the US probe will be moved toward anterior axillary line till pectoralis minor and serratus anterior muscles will be identified at 4th rib at the level of thoraco-acromial artery then the needle will be inserted in plane with the probe from caudal to cranial in an inclined way, 15mL of bupivacaine 0.25% after negative aspiration will be put into the potential space between pectoralis minor muscle and serratus muscle (PECS II). After 15 minutes of the block, surgical incision will be allowed. Drug packs will be prepared before commencement of the study by a pharmacist unaware of the nature of the study. Inadequate analgesia is defined as more than 20% increase in mean blood pressure and/or heart rate after skin incision and during surgical procedure which will be managed by administration of 1 μg/kg fentanyl. The average end-tidal isoflurane, total intraoperative fentanyl dose will be recorded. In case of failure of the block patient will be excluded.At the end of the surgical procedure, anesthesia will be discontinued and neuromuscular blockade will be reversed with neostigmine(0.05 mg/kg) IV and atropine iv (0.03 mg/kg).Patients will be extubated and shifted to the post-anesthesia care unit. In postoperative anaesthesia care unit, postoperative monitoring of the hemodynamics will be undergone by a well trained nurse who will be blinded to the study and the sensory level of the block was tested using the cold test, done by a blinded physician to the nature of the study after the operation.

.Before induction of anesthesia patients will be teached how to use a 100 cm visual analog scale (VAS) 0 =''no pain" and 100 =''worst imaginable pain"). If VAS score > 4 then a rescue dose of a fentanyl 1.0 μg kg-1 i.v. bolus will be given.

The primary outcome measures will include time of performance of each technique.

The secondary outcomes will include total dose of postoperative fentanyl consumed, visual analogue scores in addition to vital signs will be assessed at 2, 6, 10, 12, 18, 24 h by an investigator blinded to the group allocation and the nature of the study. postoperative adverse events such as hypotension and respiratory depression, postoperative nausea and vomiting (PONV) which will be evaluated using a four-point numerical scale (0=no PONV, 1=mild nausea, 2=severe nausea or vomiting once, and 3=vomiting more than once). The rescue dose of ondansetron 0.1 mg kg-1 will be given i.v. if the score is 2 or more.Moreover, the time to first dose of rescue analgesic.

ELIGIBILITY:
Inclusion Criteria:

* female patients aged from 50-65 years old elective breast surgeries ASA I II

Exclusion Criteria:

* Refusal to participate inability to communicate with the investigators or hospital staff obesity (body mass index>40 kg/m2) patients undergoing bilateral surgery male patients renal insufficiency (creatinine>1.5 mg/dL) American Society of Anesthesia (ASA) III-IV patients with incomplete medical records

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — recruitment of patients is based on representation of gender identity.
Enrollment: 60 (Actual)
Dates: Start 2019-11-10 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-07-02 (Actual)

PRIMARY OUTCOMES:
time of performance of each technique | 10 to 15 minutes
  duration of performance of each technique

SECONDARY OUTCOMES:
total dose of postoperative fentanyl consumed | 24 hours after the procedure
  dose of rescue analgesic

CONTACTS AND LOCATIONS:
Overall Officials: Nahed Effat, Study Director — Ain Shams University
Locations (1):
- Ain Shams U, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
study protocol statistical analysis data analysis
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 7 months
Access Criteria: Descriptive statistics will be carried out for numerical parametric data and presented as mean±SD, whereas categorical data will be presented as number and percentage. Variables such as demographic data andcomorbidities will be compared using the χ2-test